CLINICAL TRIAL: NCT00005449
Title: Social Support and Myocardial Ischemia
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4378; R29HL056825 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; Coronary Disease

SUMMARY:
To examine the role of social support in attenuating ischemic responses to psychological stress, both in the laboratory and during daily life.

DETAILED DESCRIPTION:
BACKGROUND:

A large quantity of epidemiological data has accumulated attesting to a link between social support and the progression of cardiovascular disease in cardiac patients. One way that social support might exerts its health effects is by attenuating physiological responses to psychological stress, since these responses have been related to cardiovascular disease. Much myocardial ischemia occurring during daily life appears to be related to periods of psychological stress, and laboratory mental stress tasks have been found to induce ischemia. Thus, the incidence, severity, and duration of myocardial ischemia might be modified by changes in the social environment.

DESIGN NARRATIVE:

There are two components to the study. In the first component, the investigators are testing the hypothesis that the presence of a supportive spouse attenuates ischemic responses to psychological stress in the laboratory. Using a counterbalanced crossover, repeated measures design, patients are asked to complete a public speaking task in the laboratory in two conditions: with a spouse present; and alone. Hemodynamic, radionuclide angiographic, and catecholamine responses to the task are assessed in both conditions.

In the second component, the investigators are examining whether married patients show reduced duration of ischemia compared to unmarried patients. In addition, they plan to examine whether presence of a supportive other (spouse, or friend in the case of unmarried patients) reduces the incidence and duration of ischemia in patients during daily life activities. Patients are asked to keep a detailed diary for a two week period to ascertain patterns of daily activities. Using these diaries and in consultation with patients, the investigators are selecting a two day period during which patients have a busy and varied schedule. Patients are then asked to follow the same pattern of activities for a 48 hour period on two consecutive weeks when heart rate, and the incidence and duration of ischemia are measured. During one week their spouse, in the case of married patients, or friend, in the case of unmarried patients, is present; during the other week patients are to repeat the activities alone.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-08; Study Completion 2001-06

REFERENCES:
- [Background] Carroll D, Sheffield D. Social psychophysiology, social circumstances, and health. Ann Behav Med. 1998 Fall;20(4):333-7. doi: 10.1007/BF02886383. PMID 10234428
- [Background] Sheffield D, Kirby DS, Biles PL, Sheps DS. Comparison of perception of angina pectoris during exercise testing in African-Americans versus Caucasians. Am J Cardiol. 1999 Jan 1;83(1):106-8, A8. doi: 10.1016/s0002-9149(98)00790-5. PMID 10073794